CLINICAL TRIAL: NCT03447990
Title: Randomized, Double-blind, Placebo-controlled, Two-Part, Adaptive Design Study of Safety, Tolerability, Preliminary Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Oral Doses of MYK-491 in Patients With Stable Heart Failure With Reduced Ejection Fraction
Brief Title: v4 Study Evaluating the Safety, Tolerability and Preliminary Pharmacokinetics and Pharmacodynamics of MYK-491
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MYK-491-003
Record Dates: First submitted 2018-02-14; First posted 2018-02-27 (Actual); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Intervention Model Description: This is a a two part study. The first part is a randomized, crossover, double-blind, placebo-controlled, two cohort, sequential ascending single dose study. All patients will receive placebo and active doses of MYK-491.
  The second part is a randomized, parallel, double-blind, placebo-controlled, sequential ascending multiple dose study. All patients will receive placebo and/or active doses of MYK-491.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1/SAD and Part 2/MAD - drug (Other): Part 1/SAD: Crossover, Single ascending dose of MYK-491/placebo
  Part 2/MAD: Parallel, multiple ascending dose of MYK-491/placebo
  Interventions: Drug: MYK-491
- Part 1/SAD and Part 2/MAD - placebo (Other): Part 1/SAD: Crossover, Single ascending dose of MYK-491/placebo
  Part 2/MAD: Parallel, multiple ascending dose of MYK-491/placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MYK-491 — Single Ascending Dose and Multiple Ascending Dose of MYK-491
  Arms: Part 1/SAD and Part 2/MAD - drug
Drug: Placebo — Single Ascending Dose and Multiple Ascending Dose of placebo
  Arms: Part 1/SAD and Part 2/MAD - placebo

SUMMARY:
The purpose of this Phase 1b/2a study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of MYK-491 in patients with stable heart failure.

ELIGIBILITY:
Key Inclusion Criteria:

* Has stable chronic heart failure with reduced ejection fraction
* Has adequate acoustic windows for echocardiography

Key Exclusion Criteria:

* Any significant structural cardiac abnormalities on Screening TTE
* At Screening, symptomatic hypotension or hypertension or bradycardia.
* Routinely scheduled outpatient intravenous (IV) infusions for heart failure (e.g., inotropes, vasodilators [e.g., nesiritide], diuretics) or routinely scheduled ultrafiltration.
* Presence of protocol specified laboratory abnormalities at Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (9):
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Prism Reseach, Saint Paul, Minnesota
  - St. Louis Heart and Vascular Cardiology, St Louis, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Heart and Vascular Center, Philadelphia, Pennsylvania
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
- Hopital Europeen Georges-Pompidou, Paris, France
- Charite Research Organization, Berlin, Germany
- Netherlands (2):
  - Groningen UMC, Groningen
  - D&A Research, Sneek
- Poland (2):
  - Wojewodzki Szpital Specjalistyczny Im M Kopernika, Lodz
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Oddzial Kardiologiczny z Pododdzialem Intensywnego Nadzoru Kardiologicznego i Pododdzialem Leczenia Zaburzen Rytmu Serca, Wroclaw
- Karolinska University Hospital, Stockholm, Sweden
- Queen Elizabeth University Hospital, Glasgow, Scotland, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- SAD Cohort 1: Participants received 3 double-blinded single ascending doses in random sequence (1 placebo, Danicamtiv 175mg and Danicamtiv 350mg) in Period A, B, and C with intervals between doses ranging from 3 to 14 days. Some participants received a fourth single dose of Danicamtiv ranging between 350mg-550mg in the optional open-label period D
- SAD Cohort 2: Participants received 3 double-blinded single ascending doses in random sequence (1 placebo, Danicamtiv 400mg and Danicamtiv 500mg) in Period A, B, and C with intervals between doses ranging from 3 to 14 days
- MAD Cohort 1: Participants received single-blinded placebo twice daily for 2 days. Participants then received double-blinded Danicamtiv 75mg (fasting) twice daily for 7 days, and 2 days of monitoring following the last dose before discharge.
- MAD Cohort 2: Participants received single-blinded placebo twice daily for 2 days. Participants then received double-blinded Danicamtiv 50mg (with food) twice daily for 7 days, and 2 days of monitoring following the last dose before discharge.
- MAD Cohort 3: Participants received single-blinded placebo twice daily for 2 days. Participants then received double-blinded Danicamtiv 75mg (with food) twice daily for 7 days, and 2 days of monitoring following the last dose before discharge.
- MAD Cohort 4: Participants received single-blinded placebo twice daily for 2 days. Participants then received double-blinded Danicamtiv 100mg (with food) twice daily for 7 days, and 2 days of monitoring following the last dose before discharge.
- MAD Placebo: Participants received single-blinded placebo twice daily for 2 days. Participants then received double-blinded placebo twice daily for 7 days, and 2 days of monitoring following the last dose before discharge.
Period: Overall Study
Arm/Group | SAD Cohort 1 | SAD Cohort 2 | MAD Cohort 1 | MAD Cohort 2 | MAD Cohort 3 | MAD Cohort 4 | MAD Placebo
Started (Started = Randomized and treated) | 8 | 4 | 6 | 9 | 9 | 6 | 10
Completed Blinded Treatment Period A (Blinded treatment period A planned in SAD Cohort 1 and 2) | 8 | 4 | 0 | 0 | 0 | 0 | 0
Completed Blinded Treatment Period B (Blinded treatment period B planned in SAD Cohort 1 and 2) | 8 | 4 | 0 | 0 | 0 | 0 | 0
Completed Blinded Treatment Period C (Blinded treatment period C planned in SAD Cohort 1 and 2) | 8 | 4 | 0 | 0 | 0 | 0 | 0
Completed Optional Open-Label Treatment Period D (Optional open-label treatment period D planned in SAD Cohort 1) | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed = completed treatment) | 8 | 4 | 6 | 9 | 9 | 6 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SAD Cohort 1 | SAD Cohort 2 | MAD Cohort 1 | MAD Cohort 2 | MAD Cohort 3 | MAD Cohort 4 | MAD Placebo | Total
Number analyzed (Participants) | 8 | 4 | 6 | 9 | 9 | 6 | 10 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.1 (9.4) | 57.5 (5.07) | 62.7 (12.50) | 63.0 (9.86) | 56.8 (5.09) | 58.5 (5.36) | 58.6 (6.98) | 59.2 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 3 | 2 | 1 | 1 | 14
  Male | 5 | 3 | 3 | 6 | 7 | 5 | 9 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 4 | 6 | 9 | 9 | 6 | 9 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 1 | 3 | 1 | 2 | 0 | 3 | 16
  White | 2 | 3 | 3 | 8 | 7 | 6 | 7 | 36
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Number of participants with any grade of treatment-emergent adverse events (TEAEs) and any grade of serious adverse events (SAEs).
Time Frame: From first dose to 30 days post last dose (Up to 2 months)
Population: All treated participants per regimen dosage
Measure: Count of Participants; unit: Participants
Groups:
- SAD Cohort 1 Danicamtiv 175mg: Participants received single dose of Danicamtiv 175mg in either period A, B, or C
- SAD Cohort 1 Danicamtiv 350mg: Participants received single dose of Danicamtiv 350mg in either period A, B, C, or D
- SAD Cohort 1 Placebo: Participants received single dose of Placebo in either period A, B, or C
- SAD Cohort 1 Danicamtiv 450mg: Participants received split dose of Danicamtiv 450mg in period D
- SAD Cohort 1 Danicamtiv 525mg: Participants received single dose of Danicamtiv 525mg in period D
- SAD Cohort 1 Danicamtiv 550mg: Participants received split dose of Danicamtiv 550mg in period D
- SAD Cohort 2 Danicamtiv 400mg: Participants received split dose of Danicamtiv 400mg
- SAD Cohort 2 Danicamtiv 500mg: Participants received split dose of Danicamtiv 500mg
- SAD Cohort 2 Placebo: Participants received single dose of Placebo
- MAD Cohort 2 Danicamtiv 50mg: Participants received single-blinded placebo twice daily for 2 days. Participants then received double-blinded Danicamtiv 50mg (with food) twice daily for 7 days, and 2 days of monitoring following the last dose before discharge
- MAD Cohort 1+3 Danicamtiv 75mg: Participants received single-blinded placebo twice daily for 2 days. Participants then received double-blinded Danicamtiv 75mg twice daily for 7 days, and 2 days of monitoring following the last dose before discharge
- MAD Cohort 4 Danicamtiv 100mg: Participants received single-blinded placebo twice daily for 2 days. Participants then received double-blinded Danicamtiv 100mg (with food) twice daily for 7 days, and 2 days of monitoring following the last dose before discharge
- MAD Cohort Placebo: Participants received single-blinded placebo twice daily for 2 days. Participants then received double-blinded Placebo twice daily for 7 days, and 2 days of monitoring following the last dose before discharge
Arm/Group | SAD Cohort 1 Danicamtiv 175mg | SAD Cohort 1 Danicamtiv 350mg | SAD Cohort 1 Placebo | SAD Cohort 1 Danicamtiv 450mg | SAD Cohort 1 Danicamtiv 525mg | SAD Cohort 1 Danicamtiv 550mg | SAD Cohort 2 Danicamtiv 400mg | SAD Cohort 2 Danicamtiv 500mg | SAD Cohort 2 Placebo | MAD Cohort 2 Danicamtiv 50mg | MAD Cohort 1+3 Danicamtiv 75mg | MAD Cohort 4 Danicamtiv 100mg | MAD Cohort Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 2 | 2 | 4 | 4 | 4 | 9 | 15 | 6 | 10
Participants
  TEAEs | 2 | 5 | 3 | 0 | 0 | 1 | 3 | 0 | 0 | 7 | 6 | 4 | 4
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Participants With Change From Baseline in Electrocardiograms (ECG) Intervals - SAD Cohorts
Description: Number of participants with change from baseline in ECGs QTcF, PR, and QRS intervals. Baseline is defined as the last non-missing value prior to the corresponding period.
Time Frame: Baseline, day 1-16, 2 hours pre-dose and at 3-, 5-, 9-, 12-, 24-, and 36-hours post-dose
Population: All treated participants in SAD Cohorts per regimen dosage
Measure: Count of Participants; unit: Participants
Arm/Group | SAD Cohort 1 Danicamtiv 175mg | SAD Cohort 1 Danicamtiv 350mg | SAD Cohort 1 Placebo | SAD Cohort 1 Danicamtiv 450mg | SAD Cohort 1 Danicamtiv 525mg | SAD Cohort 1 Danicamtiv 550mg | SAD Cohort 2 Danicamtiv 400mg | SAD Cohort 2 Danicamtiv 500mg | SAD Cohort 2 Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 2 | 2 | 4 | 4 | 4
Participants
  Change in QTcF from Baseline > 30msec | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Change in QTcF from Baseline > 60msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Change in PR from baseline > 25% | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change in QRS from baseline > 25% | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Change From Baseline in Electrocardiograms (ECG) Intervals - MAD Cohorts
Description: Number of participants with change from baseline in ECGs QTcF, PR, and QRS intervals. Baseline is defined as the last non-missing value prior to first randomized dose.
Time Frame: Baseline, Day 1-16, 2 hours pre-dose and at 7-, 24-, and 48-hours post final dose
Population: All treated participants in MAD Cohorts per regimen dosage
Measure: Count of Participants; unit: Participants
Arm/Group | MAD Cohort 2 Danicamtiv 50mg | MAD Cohort 1+3 Danicamtiv 75mg | MAD Cohort 4 Danicamtiv 100mg | MAD Cohort Placebo
Number analyzed (Participants) | 9 | 15 | 6 | 10
Participants
  Change in QTcF from Baseline > 30msec | 2 | 5 | 1 | 3
  Change in QTcF from Baseline > 60msec | 0 | 0 | 1 | 1
  Change in PR from baseline > 25% | 0 | 0 | 0 | 1
  Change in QRS from baseline > 25% | 1 | 2 | 0 | 2

4. Primary Outcome: Mean Change From Baseline in Vital Signs Part 1 - SAD Cohorts
Description: Mean change from baseline in supine systolic blood pressure (SBP) and supine diastolic blood pressure (DBP) vital signs. Baseline is defined as the last non-missing value prior to the corresponding period.
Time Frame: Baseline and at 6-hours post-dose
Population: All treated participants in SAD Cohorts per regimen dosage
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SAD Cohort 1 Danicamtiv 175mg | SAD Cohort 1 Danicamtiv 350mg | SAD Cohort 1 Placebo | SAD Cohort 1 Danicamtiv 450mg | SAD Cohort 1 Danicamtiv 525mg | SAD Cohort 1 Danicamtiv 550mg | SAD Cohort 2 Danicamtiv 400mg | SAD Cohort 2 Danicamtiv 500mg | SAD Cohort 2 Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 2 | 2 | 4 | 4 | 4
mmHg
  Supine SBP | -10.13 (12.23) | -11.38 (9.90) | -1.38 (15.02) | 16.00 (NA) — SD was not calculated because of insufficient number of events | -7.00 (19.80) | -9.50 (2.12) | 2.50 (4.359) | 01.75 (15.650) | 0.00 (11.633)
  Supine DBP | -5.50 (12.14) | 9.50 (6.44) | -5.75 (13.04) | 12.00 (NA) — SD was not calculated because of insufficient number of events | -1.00 (5.66) | -4.00 (8.49) | 4.00 (9.933) | -2.25 (17.270) | -3.00 (14.674)

5. Primary Outcome: Mean Change From Baseline in Vital Signs Part 1 - MAD Cohorts
Description: Mean change from baseline in supine systolic blood pressure (SBP) and supine diastolic blood pressure (DBP) vital signs. Baseline is defined as the last non-missing value prior to first randomized dose
Time Frame: Baseline and at 6-hours post-dose
Population: Pre-specified for data to be collected by combining all treated participants with vital signs measurements in MAD Cohorts per regimen only
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- MAD Cohorts Danicamtiv: MAD cohorts at doses ranging from 50 mg to 100 mg
- MAD Cohorts Placebo: MAD cohorts with participants that received placebo
Arm/Group | MAD Cohorts Danicamtiv | MAD Cohorts Placebo
Number analyzed (Participants) | 7 | 3
mmHg
  Supine SBP | -4.86 (7.537) | -6.33 (3.215)
  Supine DBP | -3.57 (7.323) | -5.67 (3.055)

6. Primary Outcome: Mean Change From Baseline in Vital Signs Part 2 - SAD Cohorts
Description: Mean change from baseline in heart rate (HR) vital signs. Baseline is defined as the last non-missing value prior to the corresponding period.
Time Frame: Baseline and at 6-hours post-dose
Population: All treated participants in SAD Cohorts per regimen dosage
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | SAD Cohort 1 Danicamtiv 175mg | SAD Cohort 1 Danicamtiv 350mg | SAD Cohort 1 Placebo | SAD Cohort 1 Danicamtiv 450mg | SAD Cohort 1 Danicamtiv 525mg | SAD Cohort 1 Danicamtiv 550mg | SAD Cohort 2 Danicamtiv 400mg | SAD Cohort 2 Danicamtiv 500mg | SAD Cohort 2 Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 2 | 2 | 4 | 4 | 4
Beats/min | 7.13 (6.20) | -1.25 (5.75) | 3.00 (5.50) | 5.00 (NA) — SD was not calculated because of insufficient number of events | 5.50 (0.71) | -1.50 (2.12) | 3.75 (9.743) | -0.50 (5.000) | -6.50 (13.699)

7. Primary Outcome: Mean Change From Baseline in Vital Signs Part 2 - MAD Cohorts
Description: Mean change from baseline in heart rate (HR) vital signs. Baseline is defined as the last non-missing value prior to first randomized dose
Time Frame: Baseline and at 6-hours post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | MAD Cohorts Danicamtiv | MAD Cohorts Placebo
Number analyzed (Participants) | 7 | 3
Beats/min | 3.71 (2.563) | 3.33 (2.517)

8. Primary Outcome: Number of Participants With a Troponin I Increase - SAD Cohorts
Description: Number of participants with a troponin increase is defined as when one of the following conditions was met (1) if the participant's troponin I value was normal prior to dosing (≤0.03 ng/mL), an elevated level on at least one measurement after start of dosing >2×ULN for the specific assay (>0.06 ng/mL) through Day 16. (2) If the participant's troponin I value was above the ULN for the specific assay prior to dosing, an increase >0.03 ng/mL compared to baseline on at least one measurement after start of dosing through Day 16.
Time Frame: Baseline, day 1-3, 2 hours pre-dose and at 3-, 5-, 9-, 12-, 24-, and 36-hours post-dose
Population: Pre-specified for data to be collected by combining all treated participants in SAD Cohorts per regimen only
Measure: Count of Participants; unit: Participants
Groups:
- SAD Cohorts Danicamtiv: SAD cohorts at doses ranging from 175 mg to 550 mg
- SAD Cohorts Placebo: SAD cohorts with participants that received placebo
Arm/Group | SAD Cohorts Danicamtiv | SAD Cohorts Placebo
Number analyzed (Participants) | 12 | 12
Participants | 3 | 0

9. Primary Outcome: Number of Participants With a Troponin I Increase - MAD Cohorts
Description: as for outcome 8
Time Frame: Baseline, pre-dose and 7hr post dose on treatment day 1, day 2, day 5 and pre-dose and at 7-, 24-, and 48-hours post final dose
Population: Pre-specified for data to be collected by combining all treated participants in MAD Cohorts per regimen only
Measure: Count of Participants; unit: Participants
Arm/Group | MAD Cohorts Danicamtiv | MAD Cohorts Placebo
Number analyzed (Participants) | 30 | 10
Participants | 7 | 0

10. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Number of participants with clinically significant laboratory abnormalities.
Time Frame: From first dose to 30 days post last dose (Up to 2 months)
Population: Pre-specified for data to be collected by combining all treated participants per SAD and MAD Cohort only
Measure: Count of Participants; unit: Participants
Groups:
- SAD Cohorts: SAD cohorts Placebo and Danicamtiv at doses ranging from 175 mg to 550 mg
- MAD Cohorts: MAD cohorts Placebo and Danicamtiv doses ranging from 50 mg to 100 mg
Arm/Group | SAD Cohorts | MAD Cohorts
Number analyzed (Participants) | 12 | 40
Participants | 1 | 1

11. Primary Outcome: Number of Participants With Clinically Significant Physical Examinations Abnormalities
Description: Number of participants with clinically significant physical examinations abnormalities.
Time Frame: From first dose to 30 days post last dose (Up to 2 months)
Population: Pre-specified for data to be collected by combining all treated participants per SAD and MAD Cohort only
Measure: Count of Participants; unit: Participants
Arm/Group | SAD Cohorts | MAD Cohorts
Number analyzed (Participants) | 12 | 40
Participants | 0 | 0

12. Secondary Outcome: Danicamtiv Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration (Cmax) for Danicamtiv. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
Time Frame: 1 hour pre-dose and day 1-12 at 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, and 48 hours postdose
Population: All participants that received Danicamtiv with plasma concertation data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- SAD Cohort 1 Danicamtiv 350mg Period D: Participants received single dose of Danicamtiv 350mg in period D
Arm/Group | SAD Cohort 1 Danicamtiv 175mg | SAD Cohort 1 Danicamtiv 350mg | SAD Cohort 1 Danicamtiv 450mg | SAD Cohort 1 Danicamtiv 350mg Period D | SAD Cohort 1 Danicamtiv 525mg | SAD Cohort 1 Danicamtiv 550mg | SAD Cohort 2 Danicamtiv 400mg | SAD Cohort 2 Danicamtiv 500mg | MAD Cohort 2 Danicamtiv 50mg | MAD Cohort 1+3 Danicamtiv 75mg | MAD Cohort 4 Danicamtiv 100mg
Number analyzed (Participants) | 8 | 8 | 1 | 1 | 2 | 2 | 4 | 4 | 8 | 15 | 6
ng/mL | 1476.63 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 22.72 | 2655.83 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 29.47 | 4420.00 (NA) — Coefficient of variation was not calculated because of insufficient number of events | 3590.00 (NA) — Coefficient of variation was not calculated because of insufficient number of events | 2718.51 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 4.68 | 5263.71 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 9.28 | 5337.58 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 24.65 | 5740.50 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 25.86 | 792.5 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 20.2 | 1174.3 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 19.1 | 1452.8 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 21.9

13. Secondary Outcome: Danicamtiv Time of Maximum Observed Plasma Concentration (Tmax)
Description: Time of maximum observed plasma concentration (Tmax) for Danicamtiv.
Time Frame: 1 hour pre-dose and day 1-12 at 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, and 48 hours postdose
Population: All participants that received Danicamtiv with plasma concertation data
Measure: Median (Full Range); unit: hours
Arm/Group | SAD Cohort 1 Danicamtiv 175mg | SAD Cohort 1 Danicamtiv 350mg | SAD Cohort 1 Danicamtiv 450mg | SAD Cohort 1 Danicamtiv 350mg Period D | SAD Cohort 1 Danicamtiv 525mg | SAD Cohort 1 Danicamtiv 550mg | SAD Cohort 2 Danicamtiv 400mg | SAD Cohort 2 Danicamtiv 500mg | MAD Cohort 2 Danicamtiv 50mg | MAD Cohort 1+3 Danicamtiv 75mg | MAD Cohort 4 Danicamtiv 100mg
Number analyzed (Participants) | 8 | 8 | 1 | 1 | 2 | 2 | 4 | 4 | 8 | 15 | 6
hours | 5.14 [2.0 to 6.3] | 6.18 [3.7 to 9.1] | 12.0 [12.0 to 12.0] | 4.1 [4.1 to 4.1] | 5.74 [5.4 to 6.1] | 8.93 [7.9 to 9.9] | 9.13 [6.0 to 12.2] | 9.08 [6.0 to 10.0] | 4.983 [3.00 to 9.00] | 4.000 [1.00 to 12.05] | 3.500 [2.03 to 9.00]

14. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC)
Description: Area under the plasma concentration-time curve (AUC) for Danicamtiv including the following time points: (AUC(0-12))=from time 0 to 12 hours; (AUC(0-24))=from time 0 to 24 hours; (AUC(0-48))=from time 0 to 48 hours; (AUClast)=from time 0 up to the last measurable concentration; (AUC(0-∞))=from time 0 to infinity. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
Time Frame: 1 hour pre-dose and day 1-12 at 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, and 48 hours postdose
Population: All participants that received Danicamtiv with plasma concertation data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr x ng/mL
Arm/Group | SAD Cohort 1 Danicamtiv 175mg | SAD Cohort 1 Danicamtiv 350mg | SAD Cohort 1 Danicamtiv 450mg | SAD Cohort 1 Danicamtiv 350mg Period D | SAD Cohort 1 Danicamtiv 525mg | SAD Cohort 1 Danicamtiv 550mg | SAD Cohort 2 Danicamtiv 400mg | SAD Cohort 2 Danicamtiv 500mg | MAD Cohort 2 Danicamtiv 50mg | MAD Cohort 1+3 Danicamtiv 75mg | MAD Cohort 4 Danicamtiv 100mg
Number analyzed (Participants) | 8 | 8 | 1 | 1 | 2 | 2 | 4 | 4 | 8 | 15 | 6
hr x ng/mL
  (AUC(0-12)): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 15 | 6
  (AUC(0-12)) |  |  |  |  |  |  |  |  | 7169.245 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 18.6 | 10310.794 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 20.4 | 12728.956 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 16.8
  (AUC(0-24)): number analyzed (Participants) | 8 | 8 | 1 | 1 | 2 | 2 | 4 | 4 | 0 | 0 | 0
  (AUC(0-24)) | 26411.97 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 21.31 | 48981.93 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 27.15 | 79175.02 (NA) — Coefficient of variation was not calculated because of insufficient number of events | 70138.66 (NA) — Coefficient of variation was not calculated because of insufficient number of events | 54004.82 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 4.58 | 97640.90 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 10.10 | 86110.51 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 17.56 | 97656.38 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 15.82 |  |  |
  (AUC(0-48)): number analyzed (Participants) | 8 | 8 | 1 | 1 | 2 | 2 | 4 | 4 | 0 | 0 | 0
  (AUC(0-48)) | 40068.47 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 20.91 | 76497.78 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 27.81 | 143543.52 (NA) — Coefficient of variation was not calculated because of insufficient number of events | 89356.54 (NA) — Coefficient of variation was not calculated because of insufficient number of events | 89341.77 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 2.23 | 159193.47 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 14.28 | 135385.91 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 12.21 | 161073.09 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 4.99 |  |  |
  (AUC last): number analyzed (Participants) | 8 | 8 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0
  (AUC last) | 46750.66 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 21.87 | 89216.40 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 28.49 | 182804.71 (NA) — Coefficient of variation was not calculated because of insufficient number of events | 104060.46 (NA) — Coefficient of variation was not calculated because of insufficient number of events | 106987.30 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 3.02 | 188544.49 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 16.28 |  |  |  |  |
  (AUC(0-∞)): number analyzed (Participants) | 8 | 8 | 1 | 0 | 2 | 2 | 4 | 4 | 0 | 0 | 0
  (AUC(0-∞)) | 52467.20 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 24.00 | 99576.37 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 29.22 | 234888.37 (NA) — Coefficient of variation was not calculated because of insufficient number of events |  | 126374.56 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 16.01 | 211928.81 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 16.99 | 187776.56 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 23.32 | 225087.02 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 28.27 |  |  |

15. Secondary Outcome: Apparent First-order Terminal Elimination Half-life (t1/2)
Description: Apparent first-order terminal elimination half-life (t1/2).
Time Frame: 1 hour pre-dose and day 1-12 at 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, and 48 hours postdose
Population: All participants that received Danicamtiv with plasma concertation data
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SAD Cohort 1 Danicamtiv 175mg | SAD Cohort 1 Danicamtiv 350mg | SAD Cohort 1 Danicamtiv 450mg | SAD Cohort 1 Danicamtiv 350mg Period D | SAD Cohort 1 Danicamtiv 525mg | SAD Cohort 1 Danicamtiv 550mg | SAD Cohort 2 Danicamtiv 400mg | SAD Cohort 2 Danicamtiv 500mg | MAD Cohort 2 Danicamtiv 50mg | MAD Cohort 1+3 Danicamtiv 75mg | MAD Cohort 4 Danicamtiv 100mg
Number analyzed (Participants) | 8 | 8 | 1 | 0 | 2 | 2 | 4 | 4 | 8 | 13 | 6
hours | 21.96 (4.40) | 20.95 (3.23) | 30.62 (NA) — SD was not calculated because of insufficient number of events |  | 24.73 (10.76) | 21.45 (0.30) | 24.45 (11.363) | 24.30 (13.987) | 24.466 (5.8911) | 20.573 (6.1033) | 23.319 (3.5903)

16. Secondary Outcome: Danicamtiv Accumulation Ratio for Maximum Observed Plasma Concentration AR(Cmax) - MAD Cohorts
Description: Accumulation ratio for maximum observed plasma concentration AR(Cmax) for Danicamtiv. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
Time Frame: 1 hour pre-dose and day 1-12 at 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, and 48 hours postdose
Population: All participants in MAD Cohorts that received Danicamtiv with plasma concertation data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MAD Cohort 2 Danicamtiv 50mg | MAD Cohort 1+3 Danicamtiv 75mg | MAD Cohort 4 Danicamtiv 100mg
Number analyzed (Participants) | 8 | 14 | 6
ng/mL | 3.451 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 28.0 | 3.241 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 30.2 | 3.827 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 20.6

17. Secondary Outcome: Accumulation Ratio for Area Under the Plasma Concentration-Time Curve From Time 0 to 12 Hours AR(AUC(0-12)) - MAD Cohorts
Description: Accumulation ratio for area under the plasma concentration-time curve from time 0 to 12 hours AR(AUC(0-12)) for Danicamtiv. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
Time Frame: 1 hour pre-dose and day 1-12 at 1, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, and 48 hours postdose
Population: All participants in MAD Cohorts that received Danicamtiv with plasma concertation data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr x ng/mL
Arm/Group | MAD Cohort 2 Danicamtiv 50mg | MAD Cohort 1+3 Danicamtiv 75mg | MAD Cohort 4 Danicamtiv 100mg
Number analyzed (Participants) | 8 | 14 | 6
hr x ng/mL | 3.983 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 26.5 | 3.696 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 36.4 | 4.607 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 16.5

18. Secondary Outcome: Mean Change From Baseline in Transthoracic Echocardiogram (TTE) Parameter 1 - SAD Cohorts
Description: Mean change from baseline in TTE parameter systolic ejection time (SET) according to Danicamtiv plasma concentration ranges. Baseline is defined as the last non-missing value prior to the corresponding period. Reporting arms are not mutually exclusive
Time Frame: Baseline, predose and at 3, 6, 9, and 24 hours post dose
Population: All treated participants in SAD Cohorts per Danicamtiv plasma concentration ranges (Reporting arms are not mutually exclusive)
Measure: Mean (Standard Error); unit: msec
Groups:
- SAD Cohorts <2000 ng/mL: SAD Cohorts with plasma concentration less than 2000 ng/mL
- SAD Cohorts ≥2000 ng/mL: SAD Cohorts with plasma concentration greater than or equal to 2000 ng/mL
Arm/Group | SAD Cohorts <2000 ng/mL | SAD Cohorts ≥2000 ng/mL
Number analyzed (Participants) | 7 | 12
msec | 8.04 (10.03) | 36.3 (8.2)

19. Secondary Outcome: Mean Change From Baseline in Transthoracic Echocardiogram (TTE) Parameter 2 - SAD Cohorts
Description: Mean change from baseline in TTE parameter left ventricular stroke volume (LVSV) according to Danicamtiv plasma concentration ranges. Baseline is defined as the last non-missing value prior to the corresponding period. Reporting arms are not mutually exclusive
Time Frame: Baseline, predose and at 3, 6, 9, and 24 hours post dose
Population: as for outcome 18
Measure: Mean (Standard Error); unit: mL
Arm/Group | SAD Cohorts <2000 ng/mL | SAD Cohorts ≥2000 ng/mL
Number analyzed (Participants) | 7 | 12
mL | 1.01 (3.67) | 9.01 (2.99)

20. Secondary Outcome: Mean Change From Baseline in Transthoracic Echocardiogram (TTE) Parameter 3 - SAD Cohorts
Description: Mean change from baseline in TTE parameter left ventricular ejection fraction (LVEF) and left ventricular fractional shortening (LVFS) according to Danicamtiv plasma concentration ranges. Baseline is defined as the last non-missing value prior to the corresponding period. Reporting arms are not mutually exclusive
Time Frame: Baseline, predose and at 3, 6, 9, and 24 hours post dose
Population: as for outcome 18
Measure: Mean (Standard Error); unit: Percentage of blood pumped from LV
Arm/Group | SAD Cohorts <2000 ng/mL | SAD Cohorts ≥2000 ng/mL
Number analyzed (Participants) | 7 | 12
Percentage of blood pumped from LV
  LVEF | 4.06 (2.27) | 4.44 (1.86)
  LVFS | 3.14 (1.36) | 2.81 (1.12)

21. Secondary Outcome: Mean Change From Baseline in Transthoracic Echocardiogram (TTE) Parameter 1 - MAD Cohorts
Description: Mean change from baseline in TTE parameter systolic ejection time (SET) according to Danicamtiv plasma concentration ranges. Baseline is defined as the last non-missing value prior to first randomized dose. Reporting arms are not mutually exclusive
Time Frame: Baseline, predose, and at 7 hours post dose on day 1,2,3, 4, 7, 9, 10, and 11
Population: All treated participants in MAD Cohorts per Danicamtiv plasma concentration ranges (Reporting arms are not mutually exclusive)
Measure: Mean (Standard Error); unit: msec
Groups:
- MAD Cohorts <2000 ng/mL: MAD Cohorts with plasma concentration less than 2000 ng/mL
- MAD Cohorts 2000-<3500 ng/mL: MAD Cohorts with plasma concentration between 2000 (inclusive) to 3500 (non-inclusive) ng/mL
- MAD Cohorts ≥3500 ng/mL: MAD Cohorts with plasma concentration greater than or equal to 3500 ng/mL
Arm/Group | MAD Cohorts <2000 ng/mL | MAD Cohorts 2000-<3500 ng/mL | MAD Cohorts ≥3500 ng/mL
Number analyzed (Participants) | 30 | 26 | 13
msec | 15.1 (3.51) | 35.6 (3.78) | 48.3 (4.68)

22. Secondary Outcome: Mean Change From Baseline in Transthoracic Echocardiogram (TTE) Parameter 2 - MAD Cohorts
Description: Mean change from baseline in TTE parameter left ventricular stroke volume (LVSV) according to Danicamtiv plasma concentration ranges. Baseline is defined as the last non-missing value prior to first randomized dose. Reporting arms are not mutually exclusive
Time Frame: Baseline, predose, and at 7 hours post dose on day 1,2,3, 4, 7, 9, 10, and 11
Population: as for outcome 21
Measure: Mean (Standard Error); unit: mL
Arm/Group | MAD Cohorts <2000 ng/mL | MAD Cohorts 2000-<3500 ng/mL | MAD Cohorts ≥3500 ng/mL
Number analyzed (Participants) | 30 | 26 | 13
mL | 3.126 (1.8348) | 7.843 (1.9511) | 5.685 (2.4988)

23. Secondary Outcome: Mean Change From Baseline in Transthoracic Echocardiogram (TTE) Parameter 3 - MAD Cohorts
Description: Mean change from baseline in TTE parameter left ventricular ejection fraction (LVEF) and left ventricular fractional shortening (LVFS) according to Danicamtiv plasma concentration ranges. Baseline is defined as the last non-missing value prior to first randomized dose. Reporting arms are not mutually exclusive
Time Frame: Baseline, predose, and at 7 hours post dose on day 1,2,3, 4, 7, 9, 10, and 11
Population: as for outcome 21
Measure: Mean (Standard Error); unit: Percentage of blood pumped from LV
Arm/Group | MAD Cohorts <2000 ng/mL | MAD Cohorts 2000-<3500 ng/mL | MAD Cohorts ≥3500 ng/mL
Number analyzed (Participants) | 30 | 26 | 13
Percentage of blood pumped from LV
  LVEF | -0.25 (0.872) | 1.12 (0.928) | 2.29 (1.158)
  LVFS | 0.46 (0.537) | 0.78 (0.574) | 0.51 (0.725)

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were monitored from first dose to 30 days post last dose (Up to 2 months). Participants were assessed for All-cause mortality from their date of randomization to study completion (Up to approximately 20 months)
Groups:
- SAD Cohort 1 Danicamtiv Optional Period D: Participants received Danicamtiv at either 450mg, 525mg or 550mg in period D
- MAD Cohort 1 Danicamtiv 75mg; MAD Cohort 3 Danicamtiv 75mg: Participants received single-blinded placebo twice daily for 2 days. Participants then received double-blinded Danicamtiv 75mg twice daily for 7 days, and 2 days of monitoring following the last dose before discharge
- MAD Cohort 1 Placebo; MAD Cohort 2 Placebo; MAD Cohort 3 Placebo; MAD Cohort 4 Placebo: Participants received single-blinded placebo twice daily for 2 days. Participants then received double-blinded Placebo twice daily for 7 days, and 2 days of monitoring following the last dose before discharge
Arm/Group | SAD Cohort 1 Danicamtiv 175mg | SAD Cohort 1 Danicamtiv 350mg | SAD Cohort 1 Placebo | SAD Cohort 1 Danicamtiv Optional Period D | SAD Cohort 2 Danicamtiv 400mg | SAD Cohort 2 Danicamtiv 500mg | SAD Cohort 2 Placebo | MAD Cohort 1 Danicamtiv 75mg | MAD Cohort 1 Placebo | MAD Cohort 2 Danicamtiv 50mg | MAD Cohort 2 Placebo | MAD Cohort 3 Danicamtiv 75mg | MAD Cohort 3 Placebo | MAD Cohort 4 Danicamtiv 100mg | MAD Cohort 4 Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/6 | 0/4 | 0/4 | 0/4 | 0/6 | 0/2 | 0/9 | 0/3 | 0/9 | 0/3 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/6 | 0/4 | 0/4 | 0/4 | 1/6 | 0/2 | 0/9 | 0/3 | 0/9 | 0/3 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 3/8 | 5/8 | 3/8 | 1/6 | 3/4 | 0/4 | 0/4 | 2/6 | 0/2 | 7/9 | 1/3 | 6/9 | 1/3 | 5/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAD Cohort 1 Danicamtiv 175mg (N=8) | SAD Cohort 1 Danicamtiv 350mg (N=8) | SAD Cohort 1 Placebo (N=8) | SAD Cohort 1 Danicamtiv Optional Period D (N=6) | SAD Cohort 2 Danicamtiv 400mg (N=4) | SAD Cohort 2 Danicamtiv 500mg (N=4) | SAD Cohort 2 Placebo (N=4) | MAD Cohort 1 Danicamtiv 75mg (N=6) | MAD Cohort 1 Placebo (N=2) | MAD Cohort 2 Danicamtiv 50mg (N=9) | MAD Cohort 2 Placebo (N=3) | MAD Cohort 3 Danicamtiv 75mg (N=9) | MAD Cohort 3 Placebo (N=3) | MAD Cohort 4 Danicamtiv 100mg (N=6) | MAD Cohort 4 Placebo (N=2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3.3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAD Cohort 1 Danicamtiv 175mg (N=8) | SAD Cohort 1 Danicamtiv 350mg (N=8) | SAD Cohort 1 Placebo (N=8) | SAD Cohort 1 Danicamtiv Optional Period D (N=6) | SAD Cohort 2 Danicamtiv 400mg (N=4) | SAD Cohort 2 Danicamtiv 500mg (N=4) | SAD Cohort 2 Placebo (N=4) | MAD Cohort 1 Danicamtiv 75mg (N=6) | MAD Cohort 1 Placebo (N=2) | MAD Cohort 2 Danicamtiv 50mg (N=9) | MAD Cohort 2 Placebo (N=3) | MAD Cohort 3 Danicamtiv 75mg (N=9) | MAD Cohort 3 Placebo (N=3) | MAD Cohort 4 Danicamtiv 100mg (N=6) | MAD Cohort 4 Placebo (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cardiac discomfort (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral contusion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site erosion (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Infusion site discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QRS complex prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT03447990/Prot_SAP_000.pdf